CLINICAL TRIAL: NCT07269366
Title: Surgical Versus Percutaneous Revascularization in Patients With Reduced Left Ventricular Function
Brief Title: Surgical Versus Percutaneous Revascularization in Patients With Reduced Left Ventricular Function (STICH 3.0-NL)
Acronym: STICH 3*0-NL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-009839; 01-001-2024-0545 (Other Grant/Funding Number: Dutch Heart Foundation (Hartstichting))
Record Dates: First submitted 2025-11-20; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Coronary Artery Disease (CAD); Multivessel Coronary Artery Disease; CABG; CABG in Low EF; Heart Failure; PCI; Revascularization
Keywords: coronary artery; coronary artery disease; heart failure; low ejection fraction; hfref; cabg; coronary artery bypass graft; pci; revascularization
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG (surgery) (Experimental): Patients randomized to CABG will receive CABG - aiming for full revascularization
  Interventions: Procedure: CABG
- PCI (percutaneous) (Other): Patients randomized to PCI will receive PCI - aiming for full revascularization
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: CABG — CABG (coronary artery bypass grafting)
  Arms: CABG (surgery)
Procedure: PCI — PCI (percutaneous coronary intervention)
  Arms: PCI (percutaneous)

SUMMARY:
This randomized multicenter trial compares coronary artery bypass grafting (CABG) with percutaneous coronary intervention (PCI) in 358 patients with ischemic left ventricular dysfunction and multivessel coronary disease. The study evaluates differences in survival, major cardiovascular events, and quality of life over 4 years, and contributes to the international STICH 3.0 collaboration assessing long-term outcomes.

DETAILED DESCRIPTION:
Patients with ischemic left ventricular systolic dysfunction (iLVSD) and multivessel coronary artery disease (CAD) have a poor prognosis. Coronary artery bypass grafting (CABG) has been shown to improve long-term survival in this population compared to medical therapy alone. However, CABG carries higher short-term risks, leading to underutilization in older and comorbid patients. In contrast, percutaneous coronary intervention (PCI) is frequently performed due to perceived lower procedural risk, despite limited evidence supporting its benefit in patients with LV dysfunction. Previous studies comparing PCI with medical therapy excluded patients with clear indications for revascularization, such as those with significant angina or recent acute coronary syndrome, leaving uncertainty about the optimal treatment strategy.

The STICH 3.0-NL trial is a prospective, randomized, controlled, open-label, multicenter study designed to compare CABG and PCI in patients with iLVSD (LVEF <40%) and multivessel CAD who are candidates for coronary revascularization. A total of 358 patients will be enrolled and randomized in a 1:1 ratio to undergo CABG or PCI, aiming for full revascularization.

The primary endpoint is a hierarchical composite of all-cause mortality, recurrent major adverse cardiovascular events (MACE: non-procedural myocardial infarction, stroke, or unplanned revascularization), and recurrent hospitalizations for heart failure at 4 years. Secondary endpoints include the individual components of the primary endpoint, cardiovascular mortality, periprocedural myocardial infarction, target vessel and lesion revascularization, changes in quality of life (Seattle Angina Questionnaire and KCCQ), and cost-effectiveness expressed as QALY and ICER.

The STICH 3.0-NL trial will contribute approximately 10% of the total cohort to the international STICH 3.0 collaboration, enabling long-term analyses of all-cause mortality at 5 and 10 years and providing critical evidence to guide revascularization strategies in patients with ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* LVEF≤ 40%
* Angina pectoris, CCS≥2 and/or hospitalization for ACS or heart failure within 1 year prior to randomization
* Multivessel CAD (2-3 vessel-disease with coronary lesions >70% and involvement of proximal LAD, and/or LM stenosis of >50%). Target vessels are determined by the local Heart Time
* Clinical and angiographical characteristics suitable for isolated coronary revascularization both by CABG or PCI according to the judgment of the local Heart Team
* Written informed consent

Exclusion Criteria:

* ACS < 48 hours before randomization
* Valvular/structural heart disease requiring intervention
* Contra-indications to DAPT
* Non-cardiac condition with life expectancy < 1 year
* Previous CABG
* Decompensated HF at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2034-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite of all-cause mortality, major adverse cardiovascular events, and heart failure hospitalizations | 4 years
  Outcomes will be analyzed using a hierarchical (win ratio / Finkelstein-Schoenfeld) approach to account for clinical severity

SECONDARY OUTCOMES:
Individual components of the primary endpoint | 4 years
  Analysis of each component of the primary endpoint separately - all-cause mortality, non-procedural myocardial infarction, stroke, unplanned revascularization, and heart failure hospitalizations.
Cardiovascular mortality | 4 years
  Death due to cardiovascular causes
Periprocedural myocardial infarction | Within 30 days post-procedure
  Myocardial infarction occurring during or within 30 days after the index revascularization procedure.
Target vessel and target lesion revascularization | 4 years
  Any repeat revascularization of the initially treated coronary vessel or lesion.
Change in quality of life - Kansas City Cardiomyopathy Questionnaire | at 1 and 4 years (compared to baseline)
  Change in patient-reported quality of life assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ). The KCCQ is scored 0-100 per domain, with higher scores indicating better health status. A positive change from baseline reflects improvement. A ≥5-point change is considered clinically meaningful.
Changes in quality of life - Seattle Angina Questionnaire | at 1 and 4 years (compared to baseline)
  Change in patient-reported quality of life assessed using the Seattle Angina Questionnaire (SAQ). The SAQ is scored in 5 domains from 0-100 per domain, with higher scores indicating fewer symptoms and better health status. A change of ≥5 points is generally considered clinically meaningful.
Cost-effectiveness | 4 years
  Cost-effectiveness analysis comparing CABG and PCI, expressed as quality-adjusted life years (QALY) and incremental cost-effectiveness ratio (ICER).

CONTACTS AND LOCATIONS:
Overall Officials: Erik Lipsic, Dr, Principal Investigator — University Medical Center Groningen

IPD SHARING:
Plan to Share IPD: Undecided